CLINICAL TRIAL: NCT05751538
Title: Artificial Intelligence Based on Machine Learning in Computed Tomography for Quantifying Lung Changes of Bronchiectasis Patients
Brief Title: Artificial Intelligence in Computed Tomography for Quantifying Lung Changes of Bronchiectasis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AI-BE
Record Dates: First submitted 2023-02-08; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-11

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Machine Learning; Artificial Intelligence
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Train dataset: This group is dedicated to developing an automated algorithm.
  Interventions: Other: No intervention
- Test dataset: This group is dedicated to testing the performance of an automated algorithm.
  Interventions: Other: No intervention
- Clinical Validation: This group is dedicated to assessing the clinical validity of the measurement in an independent validation cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Bronchiectasis is a chronic respiratory disease characterized by permanent bronchiectasis.The incidence and prevalence of bronchiectasis have assumed continuously grows in global. Chest computed tomography (CT) remains the imaging standard for demonstrating cystic fibrosis (CF) airway structural disease in vivo. However, visual scoring systems as an outcome measure are time consuming, require training and lack high reproducibility. Our objective was to validate a fully automated artificial intelligence (AI)-driven scoring system of CF lung disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bronchiectasis (according to the Chinese consensus, patient's previous chest CT examination must show bronchiectasis)

Exclusion Criteria:

* Patients with CT data and medical records missing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bronchiectasis and clinical examination, pulmonary function test, and CT data
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlations of the artificial intelligence-driven scores with manual scores | From date of inclusion until the date of final quantification, assessed up to 12 months
  Correlations and comparisons of the artificial intelligence-driven scores with manual scores by thoracic radiologists on CT scans of bronchiectasis patients.

SECONDARY OUTCOMES:
Correlation of the artificial intelligence-driven scores with pulmonary function test | From date of inclusion until the date of final quantification, assessed up to 12 months
  Correlation of quantitative measurement with pulmonary function

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China